CLINICAL TRIAL: NCT06814249
Title: A Prospective Cohort Study on Ligation of Pancreatic Stump With Quantified Force During Distal Pancreatectomy
Brief Title: A Prospective Cohort Study on Ligation of Pancreatic Stump After Distal Pancreatectomy
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PS-PF
Record Dates: First submitted 2024-12-20; First posted 2025-02-07 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2024-10

CONDITIONS: Distal Pancreatectomy; Postoperative Pancreatic Fistula
Keywords: Pancreatic surgery; Distal pancreatectomy; Pancreatic texture; Pancreatic stump ligation; Postoperative pancreatic fistula

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): After severing the pancreas, the pancreas was ligated at 5 mm from the pancreatic stump with a quantified force.
  Interventions: Other: ligation of pancreatic stump with a quantified force
- Control group (Active Comparator): Handle the pancreatic stump according to conventional methods (manual suturing or stapling closure).
  Interventions: Other: Manual suturing or stapling closure.

INTERVENTIONS:
Other: ligation of pancreatic stump with a quantified force — After severing the pancreas, the pancreas was ligated at 5 mm from the pancreatic stump with a quantified force.
  Arms: Experimental group
Other: Manual suturing or stapling closure. — Handle the pancreatic stump according to conventional methods (manual suturing or stapling closure).
  Arms: Control group

SUMMARY:
The goal of this clinical trial is to learn if igation of pancreatic stump with quantified force works in decrease postoperative pancreatic fistula following distal pancreatectomy. The main outcome measures are:

Postoperative pancreatic fistula; Postoperative hospital stay.

Researchers will compare ligation to other pancreatic stump closure techniques to see if it decrease postoperative pancreatic fistula and postoperative hospital stay following distal pancreatectomy.

DETAILED DESCRIPTION:
Introduction The closure of pancreatic stump after distal pancreatectomy remains controversial. Currently, the main methods of pancreatic stump closure include manual suturing and stapler closure. However, both methods carry a high risk of pancreatic fistula, which may be associated with the difficulty of balancing the provision of sufficient pancreatic duct burst pressure and ensuring blood supply to the stump. Through in vitro experiments, we demonstrated that applying quantified ligation forces to pancreatic stumps can provide a pancreatic duct burst pressure of approximately 50-70 mmHg. This burst pressure is higher than the upper limit of normal pancreatic duct pressure and lower than the normal mean arterial pressure, theoretically balancing the pancreatic duct burst pressure and stump blood supply. Therefore, we designed this prospective cohort study to verify the above hypothesis.

Methods and analysis This is a prospective cohort study at single centre in China. The major eligibility criterion is the presence of lesions planned for distal pancreatectomy. The texture of the pancreas was determined by the surgeon and the first assistant during the operation as soft, medium, or hard. After severing the pancreas, the pancreas was ligated at 5 mm from the pancreatic stump with a quantified force. Postoperative regular follow-up will be performed. The primary outcomes included pancreatic fistula and postoperative hospital stay, and the secondary outcomes included intra-abdominal infection, incision infection, and postoperative treatment costs. The primary outcomes and secondary outcomes of patients in this cohort will be statistically compared with historical data using appropriate tests.

Ethics and dissemination The study has been approved by the Ethics Committee of Union Hospital, Tongji Medical College, Huazhong University of Science and Technology(2024-0833-02). The results of the study will be published in an international peer-reviewed journal.

ELIGIBILITY:
Inclusion Criteria:

* Patients fully understand this study, voluntarily participate, and sign the Informed Consent Form (ICF);
* Age between 18 and 75 years old;
* Planned for distal pancreatectomy (including body and tail of the pancreas);
* The intended pancreatic transection line is located on the left side of the portal vein.

Exclusion Criteria:

* History of previous pancreatic surgery;
* Additional surgical procedures required for the residual pancreas;
* Proximal pancreatic duct obstruction, with planned anastomosis between the residual pancreas and the digestive tract;
* Use of long-acting somatostatin analogues during the perioperative period;
* Patients who are judged by the investigator to be unsuitable for participation in this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-11-21 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Pancreatic fistula | Up to half a year from enrollment
  Postoperative pancreatic fistula adopts the definition proposed by the International Study Group of Pancreatic Surgery.
Postoperative hospital stay | Up to half a year from enrollment
  Stay from operation to discharge.

SECONDARY OUTCOMES:
Intra-abdominal infection | Up to half a year from enrollment
  Intra-abdominal infection is evaluated based on Common Terminology Criteria for Adverse Event (CTCAE) V.5.0.
Incision infection | Up to half a year from enrollment
  Incision infection is evaluated based on Common Terminology Criteria for Adverse Event (CTCAE) V.5.0.
Postoperative treatment costs | Up to half a year from enrollment
  Treatment costs of postoperative period.

CONTACTS AND LOCATIONS:
Overall Officials: Shanmiao Gou, MD, Ph.D, Principal Investigator — Union Hospital, HUST, Wuhan, China
Locations (1):
- Uion Hospital, Tongji Medical College, HUST, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kaneda Y, Kimura Y, Saito A, Ae R, Kawahira H, Sata N. Pancreas Ligation Device for Distal Pancreatectomy: An Ex Vivo Follow-Up Porcine Study. Cureus. 2023 Sep 6;15(9):e44771. doi: 10.7759/cureus.44771. eCollection 2023 Sep. PMID 37692176
- [Background] Funamizu N, Sogabe K, Shine M, Honjo M, Sakamoto A, Nishi Y, Matsui T, Uraoka M, Nagaoka T, Iwata M, Ito C, Tamura K, Sakamoto K, Ogawa K, Takada Y. Association between the Preoperative C-Reactive Protein-to-Albumin Ratio and the Risk for Postoperative Pancreatic Fistula following Distal Pancreatectomy for Pancreatic Cancer. Nutrients. 2022 Dec 10;14(24):5277. doi: 10.3390/nu14245277. PMID 36558435
- [Background] Mungroop TH, van der Heijde N, Busch OR, de Hingh IH, Scheepers JJ, Dijkgraaf MG, Groot Koerkamp B, Besselink MG, van Eijck CH. Randomized clinical trial and meta-analysis of the impact of a fibrin sealant patch on pancreatic fistula after distal pancreatectomy: CPR trial. BJS Open. 2021 May 7;5(3):zrab001. doi: 10.1093/bjsopen/zrab001. PMID 34137446
- [Background] Matsuda T, Kawai C, Sakurai T. [NMR blood flow measurement and NMR angiography]. Nihon Rinsho. 1987 Jan;45(1):60-6. No abstract available. Japanese. PMID 3820687
- [Background] Abe K, Kitago M, Shinoda M, Yagi H, Abe Y, Oshima G, Hori S, Yokose T, Endo Y, Kitagawa Y. High risk pathogens and risk factors for postoperative pancreatic fistula after pancreatectomy; a retrospective case-controlled study. Int J Surg. 2020 Oct;82:136-142. doi: 10.1016/j.ijsu.2020.08.035. Epub 2020 Aug 27. PMID 32861892
- [Background] Miao Y, Lu Z, Yeo CJ, Vollmer CM Jr, Fernandez-Del Castillo C, Ghaneh P, Halloran CM, Kleeff J, de Rooij T, Werner J, Falconi M, Friess H, Zeh HJ, Izbicki JR, He J, Laukkarinen J, Dejong CH, Lillemoe KD, Conlon K, Takaori K, Gianotti L, Besselink MG, Del Chiaro M, Montorsi M, Tanaka M, Bockhorn M, Adham M, Olah A, Salvia R, Shrikhande SV, Hackert T, Shimosegawa T, Zureikat AH, Ceyhan GO, Peng Y, Wang G, Huang X, Dervenis C, Bassi C, Neoptolemos JP, Buchler MW; International Study Group of Pancreatic Surgery (ISGPS). Management of the pancreatic transection plane after left (distal) pancreatectomy: Expert consensus guidelines by the International Study Group of Pancreatic Surgery (ISGPS). Surgery. 2020 Jul;168(1):72-84. doi: 10.1016/j.surg.2020.02.018. Epub 2020 Apr 2. PMID 32249092
- [Background] Rozich NS, Morris KT, Garwe T, Sarwar Z, Landmann A, Siems CB, Jones A, Butler CS, McGaha PK, Axtman BC, Edil BH, Lees JS. Blame it on the injury: Trauma is a risk factor for pancreatic fistula following distal pancreatectomy compared with elective resection. J Trauma Acute Care Surg. 2019 Dec;87(6):1289-1300. doi: 10.1097/TA.0000000000002495. PMID 31765347
- [Background] Ratnayake CBB, Wells C, Hammond J, French JJ, Windsor JA, Pandanaboyana S. Network meta-analysis comparing techniques and outcomes of stump closure after distal pancreatectomy. Br J Surg. 2019 Nov;106(12):1580-1589. doi: 10.1002/bjs.11291. Epub 2019 Oct 18. PMID 31626341
- [Background] Nagakawa Y, Hijikata Y, Osakabe H, Matsudo T, Soya R, Sahara Y, Takishita C, Shirota T, Kobayashi N, Nakajima T, Hosokawa Y, Ishizaki T, Katsumata K, Tsuchida A. Why Does Postoperative Pancreatic Fistula Occur After Hand-sewn Parenchymal Closure and Staple Closure in Distal Pancreatectomy? Surg Laparosc Endosc Percutan Tech. 2019 Apr;29(2):e15-e19. doi: 10.1097/SLE.0000000000000604. PMID 30520812
- [Background] de Rooij T, van Hilst J, van Santvoort H, Boerma D, van den Boezem P, Daams F, van Dam R, Dejong C, van Duyn E, Dijkgraaf M, van Eijck C, Festen S, Gerhards M, Groot Koerkamp B, de Hingh I, Kazemier G, Klaase J, de Kleine R, van Laarhoven C, Luyer M, Patijn G, Steenvoorde P, Suker M, Abu Hilal M, Busch O, Besselink M; Dutch Pancreatic Cancer Group. Minimally Invasive Versus Open Distal Pancreatectomy (LEOPARD): A Multicenter Patient-blinded Randomized Controlled Trial. Ann Surg. 2019 Jan;269(1):2-9. doi: 10.1097/SLA.0000000000002979. PMID 30080726
- [Background] Ecker BL, McMillan MT, Allegrini V, Bassi C, Beane JD, Beckman RM, Behrman SW, Dickson EJ, Callery MP, Christein JD, Drebin JA, Hollis RH, House MG, Jamieson NB, Javed AA, Kent TS, Kluger MD, Kowalsky SJ, Maggino L, Malleo G, Valero V 3rd, Velu LKP, Watkins AA, Wolfgang CL, Zureikat AH, Vollmer CM Jr. Risk Factors and Mitigation Strategies for Pancreatic Fistula After Distal Pancreatectomy: Analysis of 2026 Resections From the International, Multi-institutional Distal Pancreatectomy Study Group. Ann Surg. 2019 Jan;269(1):143-149. doi: 10.1097/SLA.0000000000002491. PMID 28857813
- [Background] Chang YR, Kang JS, Jang JY, Jung WH, Kang MJ, Lee KB, Kim SW. Prediction of Pancreatic Fistula After Distal Pancreatectomy Based on Cross-Sectional Images. World J Surg. 2017 Jun;41(6):1610-1617. doi: 10.1007/s00268-017-3872-3. PMID 28091744
- [Background] Jang JY, Shin YC, Han Y, Park JS, Han HS, Hwang HK, Yoon DS, Kim JK, Yoon YS, Hwang DW, Kang CM, Lee WJ, Heo JS, Kang MJ, Chang YR, Chang J, Jung W, Kim SW. Effect of Polyglycolic Acid Mesh for Prevention of Pancreatic Fistula Following Distal Pancreatectomy: A Randomized Clinical Trial. JAMA Surg. 2017 Feb 1;152(2):150-155. doi: 10.1001/jamasurg.2016.3644. PMID 27784046
- [Background] Noorani A, Rangelova E, Del Chiaro M, Lundell LR, Ansorge C. Delayed Gastric Emptying after Pancreatic Surgery: Analysis of Factors Determinant for the Short-term Outcome. Front Surg. 2016 Apr 25;3:25. doi: 10.3389/fsurg.2016.00025. eCollection 2016. PMID 27200357
- [Background] Mendoza AS 3rd, Han HS, Ahn S, Yoon YS, Cho JY, Choi Y. Predictive factors associated with postoperative pancreatic fistula after laparoscopic distal pancreatectomy: a 10-year single-institution experience. Surg Endosc. 2016 Feb;30(2):649-656. doi: 10.1007/s00464-015-4255-1. Epub 2015 Jun 20. PMID 26091993
- [Background] Paye F, Micelli Lupinacci R, Bachellier P, Boher JM, Delpero JR; French Surgical Association (AFC). Distal pancreatectomy for pancreatic carcinoma in the era of multimodal treatment. Br J Surg. 2015 Feb;102(3):229-36. doi: 10.1002/bjs.9708. Epub 2014 Dec 22. PMID 25533421
- [Background] Okada K, Kawai M, Tani M, Hirono S, Miyazawa M, Shimizu A, Kitahata Y, Yamaue H. Isolated Roux-en-Y anastomosis of the pancreatic stump in a duct-to-mucosa fashion in patients with distal pancreatectomy with en-bloc celiac axis resection. J Hepatobiliary Pancreat Sci. 2014 Mar;21(3):193-8. doi: 10.1002/jhbp.16. Epub 2013 Jul 22. PMID 23878017
- [Background] Rostas JW, Richards WO, Thompson LW. Improved rate of pancreatic fistula after distal pancreatectomy: parenchymal division with the use of saline-coupled radiofrequency ablation. HPB (Oxford). 2012 Aug;14(8):560-4. doi: 10.1111/j.1477-2574.2012.00499.x. Epub 2012 Jun 11. PMID 22762405
- [Background] Diener MK, Seiler CM, Rossion I, Kleeff J, Glanemann M, Butturini G, Tomazic A, Bruns CJ, Busch OR, Farkas S, Belyaev O, Neoptolemos JP, Halloran C, Keck T, Niedergethmann M, Gellert K, Witzigmann H, Kollmar O, Langer P, Steger U, Neudecker J, Berrevoet F, Ganzera S, Heiss MM, Luntz SP, Bruckner T, Kieser M, Buchler MW. Efficacy of stapler versus hand-sewn closure after distal pancreatectomy (DISPACT): a randomised, controlled multicentre trial. Lancet. 2011 Apr 30;377(9776):1514-22. doi: 10.1016/S0140-6736(11)60237-7. PMID 21529927
- [Background] Ferrone CR, Warshaw AL, Rattner DW, Berger D, Zheng H, Rawal B, Rodriguez R, Thayer SP, Fernandez-del Castillo C. Pancreatic fistula rates after 462 distal pancreatectomies: staplers do not decrease fistula rates. J Gastrointest Surg. 2008 Oct;12(10):1691-7; discussion 1697-8. doi: 10.1007/s11605-008-0636-2. Epub 2008 Aug 13. PMID 18704597
- [Background] Kleeff J, Diener MK, Z'graggen K, Hinz U, Wagner M, Bachmann J, Zehetner J, Muller MW, Friess H, Buchler MW. Distal pancreatectomy: risk factors for surgical failure in 302 consecutive cases. Ann Surg. 2007 Apr;245(4):573-82. doi: 10.1097/01.sla.0000251438.43135.fb. PMID 17414606
- [Background] Okazaki K, Yamamoto Y, Ito K. Endoscopic measurement of papillary sphincter zone and pancreatic main ductal pressure in patients with chronic pancreatitis. Gastroenterology. 1986 Aug;91(2):409-18. doi: 10.1016/0016-5085(86)90576-7. PMID 3721126
- [Background] Okazaki K, Yamamoto Y, Kagiyama S, Tamura S, Sakamoto Y, Nakazawa Y, Morita M, Yamamoto Y. Pressure of papillary sphincter zone and pancreatic main duct in patients with chronic pancreatitis in the early stage. Scand J Gastroenterol. 1988 May;23(4):501-7. doi: 10.3109/00365528809093901. PMID 3381070